CLINICAL TRIAL: NCT06240065
Title: Successful Fiber Food Introduction in Short Bowel Syndrome
Acronym: GREENBEANS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Wenjing Zong, Assistant Professor in Pediatric Gastroenterology, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-1152
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Short Gut Syndrome
Keywords: nutrition; fiber; sbs; microbiome; metabolome
MeSH Terms: conditions — Short Bowel Syndrome; MYH9-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Bowel Syndrome Arm (Experimental): Patients with SBS will be initiated on green bean purees added to enteral formula recipes, based on kilocalories of enteral formula over 3 weeks. During week 1 subjects will prepare and add 50 mL green bean puree per 1000kcal of enteral feed (5%) to their formula mixture, increasing to 100ml (10%) and 150ml (15%) during weeks 2 and 3, respectively.
  Interventions: Other: Green bean puree
- Control Arm (Active Comparator): Patients without SBS will be initiated on green bean purees added to enteral formula recipes, based on kilocalories of enteral formula over 3 weeks. During week 1 subjects will prepare and add 50 mL green bean puree per 1000kcal of enteral feed (5%) to their formula mixture, increasing to 100ml (10%) and 150ml (15%) during weeks 2 and 3, respectively.
  Interventions: Other: Green bean puree

INTERVENTIONS:
Other: Green bean puree — Green bean puree as a proxy for fiber-foods

SUMMARY:
Short bowel syndrome (SBS) is a rare but challenging condition in which patients have insufficient bowel length to meet fluid, electrolyte, and nutrient requirements without parenteral support.

The purpose of this study is to determine how well dietary fiber is tolerated in patients with or without short bowel syndrome based on assessment of gastrointestinal symptoms, weight, and corresponding changes in microbiome composition and metabolomics.

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) is a rare but challenging condition in which patients have insufficient bowel length to meet fluid, electrolyte, and nutrient requirements without parenteral support. The goal of SBS treatment is to achieve enteral autonomy using strategies that optimize intestinal absorption while minimizing unpleasant gastrointestinal (GI) side effects. One strategy that has emerged is the addition of soluble fiber to enteral formula, and this strategy has gained popularity in clinical practice as fiber-rich formulas comprised of blenderized whole foods have become commercially available. However, the investigators' preliminary observations suggest that patients with SBS have variable tolerance and growth outcomes on these blenderized feeds. To date, there are no clinical studies documenting the effects of dietary fiber in SBS patients and guidance in enteral nutrition advancement is lacking in this medically complex population. The current study aims to explore the tolerance of controlled fiber addition to enteral formula based on assessment of GI symptoms, and corresponding changes in microbiome composition, and metabolomics in pediatric patients with SBS versus non-SBS controls. The investigators will use a practical approach with fiber introduction and slowly advance to goal fiber intake to understand the factors leading to continuation. Stool, urine, and plasma samples collected pre- and post- intervention will help identify biomarkers that would predict successful fiber tolerance and optimize selection of patients for fiber introduction. While there is no intent to treat, mitigate, prevent, diagnose or cure the symptoms of SBS, the study may help shed light on the underlying mechanism for intolerance to dietary fiber.

ELIGIBILITY:
Inclusion Criteria:

* Actively follows at UTSW outpatient clinics
* SBS arm specific: History of SBS diagnosis. History of short bowel syndrome based on surgical/imaging records. Small bowel is in continuity with some portion of colon
* Control arm specific: No history of intestinal pathologies
* No or negligible amount (few bites of fiber-containing foods okay) of fiber in tube feeds or by mouth at baseline
* Less than 20% calories from oral food not containing fiber while the other 80% may be by enteral and/or parenteral feedings
* At least 20% calories from fiber-free formula taken orally or via tube
* Antibiotic use is allowed, however, should be on a stable regimen of antibiotics starting from 2 weeks prior to intervention until end of study or end of week 3 whichever is sooner
* Previous history of fiber introduction failure is acceptable as long as clinically stable at the time of recruitment
* Fiber supplementation is appropriate per primary physician

Exclusion Criteria:

* SBS Arm specific: No diagnosis of SBS.
* Control Arm specific: has baseline intestinal diseases
* Small bowel and colon not in continuity (Ex: presence of ileostomy or jejunostomy)
* >5% changes in percentage of calories from PO, EN and/or PN during the intervention
* Addition/discontinuation/significant alteration to antibiotics regimen during study period
* Primary physician does not think fiber supplementation is appropriate clinically

Ages: 4 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Clinical tolerance | 3 weeks-6 months
  To assess the rate of clinical intolerance leading to discontinuation of green beans and symptoms/signs associated with discontinuation of fiber addition in SBS vs controls (no score/scale will be used)

SECONDARY OUTCOMES:
Microbiome/Metabolome Analysis | 3 weeks-6 months
  To assess the correlation between clinical tolerance of fiber and microbiome/metabolome changes in SBS vs controls

CONTACTS AND LOCATIONS:
Overall Officials: Wenjing Zong, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Children's Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided